CLINICAL TRIAL: NCT06316557
Title: HOPE From the Cerebellum: TMS-Induced Cognitive Recovery After Stroke
Acronym: HOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zi-Xiao Li (Other)
Responsible Party: Sponsor-Investigator, Zi-Xiao Li, Dr., Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-A-2022063
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Post-stroke Cognitive Impairment; Ischemic Stroke
Keywords: Post-stroke Cognitive Impairment; Repetitive transcranial magnetic stimulation; High-frequency; Cerebellar
MeSH Terms: conditions — Ischemic Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Multicenter Randomized Double-Blind Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- iTBS group (Experimental): iTBS on the contralesional cerebellum
  Interventions: Device: iTBS group
- control group (Placebo Comparator): shame stimulation on the contralesional cerebellum
  Interventions: Device: control group

INTERVENTIONS:
Device: iTBS group — iTBS on the contralesional cerebellum, twice a day for seven days
  Arms: iTBS group
Device: control group — shame stimulation on the contralesional cerebellum, twice a day for seven days
  Arms: control group

SUMMARY:
The objective of this clinical trial is to investigate the effectiveness and safety of repetitive transcranial magnetic stimulation (rTMS) in the cerebellum for individuals with post-stroke cognitive impairment. Participants will undergo rTMS in the cerebellar hemisphere opposite the lesion site, once daily for a total of five days.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to investigate the effectiveness and safety of intermittent theta burst stimulation ( iTBS) in the cerebellum for individuals with post-stroke cognitive impairment. The trial aims to answer two main questions: (1) What is the effectiveness of iTBS in improving post-stroke cognitive impairment? (2) Is iTBS in the cerebellum safe for individuals with post-stroke cognitive impairment? Participants will undergo iTBS in the cerebellar opposite the lesion site, twice daily for five days. The control group will receive sham rTMS with the same parameters and positions.

ELIGIBILITY:
Key inclusion criteria:

(1)ischemic stroke, with an initial incident occurring within 2 weeks;(2)MoCA<26;

Key exclusion criteria:

(1)Cerebral hemorrhage or subarachnoid hemorrhage;(2)A pre-existing history of epilepsy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of improving cognitive function of post-stroke cognitive impairment | 3 months follow-up after treatment
  The change of MoCA between baseline and 3 months follow-up

SECONDARY OUTCOMES:
The safety of improving cognitive function of post-stroke cognitive impairment | day1-day7
  Incidence of epilepsy during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zixiao LI, Dr., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No